CLINICAL TRIAL: NCT05052892
Title: A Novel Spleen-dedicated Stiffness Measured by FibroScan to Evaluate Cirrhotic Portal Hypertension (CHESS2105): A Prospective, Multicenter Study
Brief Title: A Novel Spleen-dedicated Stiffness Measured by FibroScan to Evaluate Cirrhotic Portal Hypertension (CHESS2105)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Shulan (Hangzhou) Hospital (Other); The Third People's Hospital of Taiyuan (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Professor, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2105
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Portal Hypertension
Keywords: cirrhosis; spleen stiffness; portal hypertension; hepatic venous pressure gradient
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Patients were fulfilled diagnosis of cirrhosis based on radiological, histological features of liver cirrhosis.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient
- Validation cohort: Patients were fulfilled diagnosis of cirrhosis based on radiological, histological features of liver cirrhosis.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient

INTERVENTIONS:
Diagnostic Test: Hepatic venous pressure gradient — All patients underwent measurement of HVPG under local anesthesia.

SUMMARY:
Portal hypertension contributed to the main complications of liver cirrhosis. Currently, hepatic venous pressure gradient (HVPG) was the reference standard for evaluating portal pressure in patients with cirrhosis. However, the practice of HVPG is limited to require the extensive experience and highly specialized centers. In recent years, non-invasive methods were proposed to predict the degree of cirrhotic portal hypertension. Of them, liver stiffness measured by FibroScan had shown good performance for predicting clinically significant portal hypertension. However, the correlation between liver stiffness and HVPG was poor when HVPG was more than 12mmHg. Since the spleen was stiffer than the liver, the current vibration-controlled transient elastography examination is dedicated to the liver, rather than the spleen. Very recently, a novel spleen-dedicated stiffness measured by FibroScan was proposed. The prospective, multicenter study aims to evaluate the correlation between SS (measured by the novel FibroScan) and HVPG, and further develop a novel model based on SS for predicting the liver decompensation in patients with compenstaed cirrhosis.

DETAILED DESCRIPTION:
Portal hypertension contributed to the main complications of liver cirrhosis. Currently, hepatic venous pressure gradient (HVPG) was the reference standard for evaluating portal pressure in patients with cirrhosis. However, the practice of HVPG is limited to require the extensive experience and highly specialized centers. In recent years, non-invasive methods were proposed to predict the degree of cirrhotic portal hypertension. Of them, liver stiffness measured by FibroScan had shown good performance for predicting clinically significant portal hypertension. However, the correlation between liver stiffness and HVPG was poor when HVPG was more than 12mmHg. Since the spleen was stiffer than the liver, the current vibration-controlled transient elastography examination is dedicated to the liver, rather than the spleen. Very recently, a novel spleen-dedicated stiffness measured by FibroScan was proposed. The prospective, multicenter study (CHESS2105 leaded by The First Hospital of Lanzhou University and Shulan (Hangzhou) Hospital) aims to evaluate the correlation between SS (measured by the novel FibroScan) and HVPG, and further develop a novel model based on SS for predicting the liver decompensation in patients with compenstaed cirrhosis.

ELIGIBILITY:
Inclusion criteria:

1. age above or equal to 18-year-old
2. fulfilled diagnosis of cirrhosis based on radiological, histological features of liver cirrhosis
3. signed informed consent

Exclusion criteria:

1. Non-cirrhotic portal hypertension
2. Lactation or pregnancy
3. Suspicious or confirmed hepatocellular carcinoma
4. Asplenia or splenectomy
5. Incomplete clinical information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients was fulfilled the diagnosis of cirrhosis based on radiological, histological features of liver cirrhosis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-28 (Estimated); Primary Completion 2025-09-27 (Estimated); Study Completion 2025-09-27 (Estimated)

PRIMARY OUTCOMES:
Accuracy of a new model based on spleen stiffness (kPa) measured by transient elastography for diagnosing portal hypertension. | 1 years
  In HVPG (mmHg) as reference method in evaluating portal pressure measured by intervention specialist , to develop a new model based on spleen stiffness (kPa) measured by transient elastography and evaluate the accuracy in diagnosing portal hypertension.

SECONDARY OUTCOMES:
Accuracy of model based on spleen stiffness (kPa) measured by transient elastography for predicting incidence of liver decompensation in patients with compenstaed cirrhosis | 3 years
  To develop a novel model based on spleen stiffness (kPa) measured by transient elastography for predicting the incidence of liver decompensation in patients with compenstaed cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, MD, Study Chair — Shulan (Hangzhou) Hospital; Xiaolong Qi, MD, Principal Investigator — LanZhou University; Huadong Yan, MD, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (3):
- China (3):
  - Shulan (Hangzhou) Hospital, Hangzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - The Third People's Hospital of Taiyuan, Taiyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Groszmann RJ, Wongcharatrawee S. The hepatic venous pressure gradient: anything worth doing should be done right. Hepatology. 2004 Feb;39(2):280-2. doi: 10.1002/hep.20062. No abstract available. PMID 14767976
- [Background] Bureau C, Metivier S, Peron JM, Selves J, Robic MA, Gourraud PA, Rouquet O, Dupuis E, Alric L, Vinel JP. Transient elastography accurately predicts presence of significant portal hypertension in patients with chronic liver disease. Aliment Pharmacol Ther. 2008 Jun;27(12):1261-8. doi: 10.1111/j.1365-2036.2008.03701.x. Epub 2008 Apr 4. PMID 18397389
- [Background] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Background] Vizzutti F, Arena U, Romanelli RG, Rega L, Foschi M, Colagrande S, Petrarca A, Moscarella S, Belli G, Zignego AL, Marra F, Laffi G, Pinzani M. Liver stiffness measurement predicts severe portal hypertension in patients with HCV-related cirrhosis. Hepatology. 2007 May;45(5):1290-7. doi: 10.1002/hep.21665. PMID 17464971
- [Background] Bastard C, Miette V, Cales P, Stefanescu H, Festi D, Sandrin L. A Novel FibroScan Examination Dedicated to Spleen Stiffness Measurement. Ultrasound Med Biol. 2018 Aug;44(8):1616-1626. doi: 10.1016/j.ultrasmedbio.2018.03.028. Epub 2018 May 3. PMID 29731186
- [Background] Stefanescu H, Marasco G, Cales P, Fraquelli M, Rosselli M, Ganne-Carrie N, de Ledinghen V, Ravaioli F, Colecchia A, Rusu C, Andreone P, Mazzella G, Festi D. A novel spleen-dedicated stiffness measurement by FibroScan(R) improves the screening of high-risk oesophageal varices. Liver Int. 2020 Jan;40(1):175-185. doi: 10.1111/liv.14228. Epub 2019 Sep 11. PMID 31444849